CLINICAL TRIAL: NCT05485805
Title: A Randomized, Double-Blind, Single-Dose, Parallel, Placebo-Controlled Pivotal Trial to Confirm the Efficacy of a Fixed Dose Combination Tablet of Naproxen Sodium and Caffeine to Effectively Alleviate Postsurgical Dental Pain
Brief Title: A Study to Learn How Well a Single Dose of the Study Treatment Naproxen Sodium and Caffeine Combined in One Tablet (Fixed-dose Combination) Works to Relieve Pain After Dental Surgeries Compared to the Single Ingredients and to Placebo
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22093; 2022-003274-22 (EudraCT Number)
Record Dates: First submitted 2022-07-28; First posted 2022-08-03 (Actual); Results first posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Postoperative Dental Pain
Keywords: Dental pain
MeSH Terms: conditions — Toothache | interventions — Naproxen; Caffeine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Naproxen sodium/caffeine - Dose 1 (Experimental): Participants will receive a single dose of one tablet of naproxen sodium/caffeine plus one tablet of placebo after extraction of third molars.
  Interventions: Drug: Naproxen sodium and caffeine (BAY2880376)
- Naproxen sodium/caffeine - Dose 2 (Experimental): Participants will receive a single dose of two tablets of naproxen sodium/caffeine after extraction of third molars.
  Interventions: Drug: Naproxen sodium and caffeine (BAY2880376)
- Naproxen sodium (Experimental): Participants will receive a single dose of one tablet of naproxen sodium plus one tablet of placebo after extraction of third molars.
  Interventions: Drug: Naproxen sodium (Aleve)
- Caffeine (Experimental): Participants will receive a single dose of two tablets of caffeine after extraction of third molars.
  Interventions: Drug: Caffeine
- Placebo (Placebo Comparator): Participants will receive a single dose of two tablets of matching placebo after extraction of third molars.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naproxen sodium and caffeine (BAY2880376) — Tablet, oral use, single dose
  Arms: Naproxen sodium/caffeine - Dose 1; Naproxen sodium/caffeine - Dose 2
Drug: Naproxen sodium (Aleve) — Tablet, oral use, single dose
  Arms: Naproxen sodium
Drug: Caffeine — Tablet, oral use, single dose
  Arms: Caffeine
Drug: Placebo — Tablet, oral use, single dose
  Arms: Placebo

SUMMARY:
Researchers are looking for a better way to relieve pain in people, such as after dental surgery.

Participants in this study, have had 3 or 4 third molars (cheek teeth) removed and subsequently have moderate to severe tooth pain.

The study treatment naproxen sodium suppresses inflammatory pain by reducing inflammation.

In the US, naproxen has been marketed since 1976, and naproxen sodium has been approved for over-the-counter (OTC) use since 1994 for the temporary relief of minor aches and pains. Caffeine, which is generally consumed as coffee, tea, or cocoa, has been shown to enhance the effect of various painkillers, and therefore is accepted as an additive.

The main purpose of this study is to learn how well a fixed-dose combination of naproxen sodium and caffeine relieves pain compared to each single ingredient as well as to placebo in participants after molar removal.

A placebo is a treatment that looks like a medicine but does not have any medicine in it.

To answer this, the researchers will compare the amount of pain decrease over 8 hours in participants who received a single dose of either:

* 1 fixed-dose tablet of naproxen sodium/caffeine
* 2 fixed-dose tablets of naproxen sodium/caffeine
* naproxen sodium only
* caffeine only
* or placebo The study participants will be randomly (by chance) assigned to one of the five treatment groups. They will take a single dose of two tablets by mouth within 4.5 hours after the surgery. If there is no pain relief within 2 hours after intake, other painkillers may be given.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, ambulatory, male or female volunteers 16 years of age or older;
* Body mass index (BMI) 18.5 to 35.0 kg/m^2 inclusive as measured by the National Institutes of Health (NIH) BMI Calculator;
* Participants will undergo surgical extraction of three or four third molars, two of which must be mandibular molars. Maxillary third molars may be removed regardless of impaction level. The mandibular extractions must have a trauma rating of mild or moderate and meet one of the following scenarios: two full bony impactions; two partial bony impactions; one full bony impaction in combination with one partial bony impaction. Supernumerary teeth present may also be removed at the discretion of the oral surgeon;
* Have not taken any form of medication, nutritional supplements with analgesic properties (e.g. gamma-Aminobutyric acid [GABA], turmeric) or herbal supplements (i.e., St. John's Wort) within 5 days of admission (except for oral contraceptives, prophylactic antibiotics, multivitamin supplements, or other routine medications to treat benign conditions (such as antibiotics to treat acne), and agree not to take any medication (other than that provided to them) throughout the study;
* Use of only short-acting local anesthetic (e.g., mepivacaine or lidocaine) preoperatively, with or without a vasoconstrictor and nitrous oxide at the discretion of the Investigator;
* Have moderate to severe postoperative pain on the Categorical Pain Intensity Scale (a score of at least 2 on a 4 point scale) and a score of ≥ 5 on the 0-10 pain intensity Numerical Rating Scale (NRS) within 4.5 hours post-surgery.

Exclusion Criteria:

* History of hypersensitivity to naproxen sodium, caffeine, ibuprofen, nonsteroidal anti-inflammatory drug (NSAIDS), aspirin, similar pharmacological agents, local anesthetics, rescue medication or components of the investigational products;
* Evidence or history of clinically significant (in the judgment of the investigator) hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular (including hypertension and cardiac arrhythmia), hepatic, psychiatric, neurologic diseases, or malignancies within the last 5 years;
* Participants with the following medical conditions may be eligible at the discretion of the investigator: attention deficit hyperactivity disorder (ADHD) on a stable dose regimen of methylphenidate/(dextro) amphetamine for at least 6 months; participants with hypothyroidism on a stable dose of synthetic thyroid hormone for at least 6 months;
* Have received any form of treatment in the form of medication for depression in the past 6 months or any form of psychotropic agent (including selective serotonin uptake inhibitors [SSRI] but excluding ADHD medications described above) within the last 6 months;
* Relevant concomitant disease such as asthma (exercise induced asthma is permitted);
* Current or past history of gastrointestinal ulceration, gastrointestinal bleeding or other bleeding disorder(s);
* Acute illness or active local infection prior to surgery that can interfere with the conduct of the study in the judgment of the investigator;
* Use of any over-the-counter (OTC) or prescription medications with which the administration of naproxen, acetaminophen, ibuprofen, any other NSAID, (e.g., tramadol) or if a medication is contraindicated;
* Use of any medications within 5 days of surgery until discharge from the study site (except oral contraceptives, prophylactic antibiotics, synthetic thyroid hormones, methylphenidate or medications to treat benign conditions such as antibiotics to treat acne);
* Use of caffeine within 2 days prior to the study;
* Habits of high consumption of caffeine (>400 mg/day equivalent to about 3-4 cups of coffee per day);
* Habituation to analgesic drugs including opioids (i.e., routine use of oral analgesics 5 or more times per week for greater than 3 weeks within the past 2 years);
* Surgeon's trauma rating of severe following surgery.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 541 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-01-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- JBR Clinical Research, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The clinical study was conducted at a single study site in the United States between 21 September 2022 (first participant first visit) and 29 January 2024 (last participant last visit).
Pre-assignment Details: A total of 750 participants were screened at a single study center in the United States. 541 participants were randomly assigned to study intervention.
Groups:
- Naproxen Sodium/ Caffeine 220/65 mg: Participants received one tablet of the fixed dose combination Naproxen sodium/Caffeine 220/65 mg and one tablet of placebo.
- Naproxen Sodium/Caffeine 2x220/65 mg: Participants received two tablets of the fixed dose combination Naproxen sodium/Caffeine 220/65 mg.
- Naproxen Sodium 220 mg: Participants received one tablet of Naproxen sodium 220 mg and one tablet of placebo.
- Caffeine 100 mg: Participants received one tablet Caffeine 100 mg one tablet of placebo.
- Placebo: Participants received two tablets of placebo.
Period: Overall Study
Arm/Group | Naproxen Sodium/ Caffeine 220/65 mg | Naproxen Sodium/Caffeine 2x220/65 mg | Naproxen Sodium 220 mg | Caffeine 100 mg | Placebo
Started | 147 | 148 | 147 | 50 | 49
Completed | 145 | 144 | 142 | 49 | 47
Not Completed | 2 | 4 | 5 | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2 | 2 | 0 | 2
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 3 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naproxen Sodium/ Caffeine 220/65 mg | Naproxen Sodium/Caffeine 2x220/65 mg | Naproxen Sodium 220 mg | Caffeine 100 mg | Placebo | Total
Number analyzed (Participants) | 147 | 148 | 147 | 50 | 49 | 541
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.3 (2.13) | 18.1 (1.99) | 18.1 (1.84) | 17.7 (1.82) | 17.9 (2.05) | 18.1 (1.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 70 | 67 | 22 | 23 | 243
  Male | 86 | 78 | 80 | 28 | 26 | 298
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 0 | 0 | 0 | 2
  Asian | 2 | 1 | 4 | 2 | 2 | 11
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 5 | 1 | 0 | 9
  Black or African American | 2 | 0 | 1 | 1 | 0 | 4
  White | 140 | 139 | 135 | 45 | 46 | 505
  More than one race | 2 | 2 | 1 | 1 | 0 | 6
  Unknown or Not Reported | 0 | 2 | 1 | 0 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Sum of Pain Intensity Difference (SPID) Over 8 Hours Post-dose
Description: Pain intensity scale is the Numerical Rating Scale measured from 0 to 10, where 0 indicates no pain and 10 means the wors pain imaginable.
  Pain intensity Difference (PID) is calculated by subtracting the pain intensity at different time points in the post-dose time point from the pain intensity at baseline.
  The summed pain intensity difference (SPID) is to be calculated by multiplying the PID score at each post dose time point by the duration (in hours) since the preceding time point and then summing the values over the relevant time period. For SPID (0-8), eight PIDs are summed up, which is minimally 0, if there is no pain relief or maximally 80, if there is very strong pain and significant pain relief.
Time Frame: Up to 8 hours post-dose
Measure: Least Squares Mean (Standard Error); unit: Points on scale
Arm/Group | Naproxen Sodium/ Caffeine 220/65 mg | Naproxen Sodium/Caffeine 2x220/65 mg | Naproxen Sodium 220 mg | Caffeine 100 mg | Placebo
Number analyzed (Participants) | 147 | 148 | 147 | 50 | 49
Points on scale | 31.293 (1.441) [lower limit 1.441] | 37.242 (1.436) [lower limit 1.436] | 31.082 (1.443) [lower limit 1.443] | 5.146 (2.470) [lower limit 2.470] | 8.622 (2.521) [lower limit 2.521]
Statistical Analysis 1: Comparison: Naproxen Sodium/ Caffeine 220/65 mg vs Naproxen Sodium/Caffeine 2x220/65 mg; Test type: Other; p = 0.004, ANCOVA; Geometric LS means = -5.95, 95% CI 2-sided [-9.946 to -1.954]
Statistical Analysis 2: Comparison: Naproxen Sodium/Caffeine 2x220/65 mg vs Naproxen Sodium 220 mg; Test type: Other; p = 0.003, ANCOVA; Geometric LS means = 6.161, 95% CI 2-sided [2.161 to 10.161]
Statistical Analysis 3: Comparison: Naproxen Sodium 220 mg vs Caffeine 100 mg; Test type: Other; p < 0.001, ANCOVA; Geometric LS means = 25.936, 95% CI 2-sided [20.317 to 31.556]
Statistical Analysis 4: Comparison: Caffeine 100 mg vs Placebo; Test type: Other; p = 0.325, ANCOVA; Geometric LS means = -3.476, 95% CI 2-sided [-10.41 to 3.457]
Statistical Analysis 5: Comparison: Naproxen Sodium/ Caffeine 220/65 mg vs Naproxen Sodium 220 mg; Test type: Other; p = 0.918, ANCOVA; Geometric LS means = 0.211, 95% CI 2-sided [-3.798 to 4.22]
Statistical Analysis 6: Comparison: Naproxen Sodium/Caffeine 2x220/65 mg vs Caffeine 100 mg; Test type: Other; p < 0.001, ANCOVA; Geometric LS means = 32.097, 95% CI 2-sided [26.484 to 37.71]
Statistical Analysis 7: Comparison: Naproxen Sodium 220 mg vs Placebo; Test type: Other; p < 0.001, ANCOVA; Geometric LS means = 22.46, 95% CI 2-sided [16.753 to 28.166]
Statistical Analysis 8: Comparison: Naproxen Sodium/ Caffeine 220/65 mg vs Caffeine 100 mg; Test type: Other; p < 0.001, ANCOVA; Geometric LS means = 26.147, 95% CI 2-sided [20.529 to 31.765]
Statistical Analysis 9: Comparison: Naproxen Sodium/Caffeine 2x220/65 mg vs Placebo; Test type: Other; p < 0.001, ANCOVA; Geometric LS means = 28.62, 95% CI 2-sided [22.921 to 34.32]
Statistical Analysis 10: Comparison: Naproxen Sodium/ Caffeine 220/65 mg vs Placebo; Test type: Other; p < 0.001, ANCOVA; Geometric LS means = 22.671, 95% CI 2-sided [16.966 to 28.375]

2. Secondary Outcome: Sum of Pain Intensity Differences From 0 to 2, 4, 6, 12 and 24 Hours Post-dose
Description: Pain intensity scale is the Numerical Rating Scale measured from 0 to 10, where 0 indicates no pain and 10 means the wors pain imaginable.
  Pain intensity Difference (PID) is calculated by subtracting the pain intensity at different time points in the post-dose time point from the pain intensity at baseline.
  The summed pain intensity difference (SPID) is to be calculated by multiplying the PID score at each post dose time point by the duration (in hours) since the preceding time point and then summing the values over the relevant time period. For SPID(0-i), i PIDs are summed up, which minimally is 0, if there is no pain relief or maximally i*10, if there is very strong pain and significant pain relief.
Time Frame: from 0 to 2, 4, 6, 12 and 24 hours post-dose
Measure: Least Squares Mean (Standard Error); unit: Points on scale
Arm/Group | Naproxen Sodium/ Caffeine 220/65 mg | Naproxen Sodium/Caffeine 2x220/65 mg | Naproxen Sodium 220 mg | Caffeine 100 mg | Placebo
Number analyzed (Participants) | 147 | 148 | 147 | 50 | 49
Points on scale
  0-2 hours post-dose | 7.347 (0.341) [lower limit 0.341] | 8.950 (0.340) [lower limit 0.340] | 7.973 (0.341) [lower limit 0.341] | 1.876 (0.585) [lower limit 0.585] | 1.567 (0.597) [lower limit 0.597]
  0-4 hours post-dose | 15.899 (0.688) [lower limit 0.688] | 19.210 (0.686) [lower limit 0.686] | 16.627 (0.689) [lower limit 0.689] | 2.924 (1.179) [lower limit 1.179] | 3.982 (1.204) [lower limit 1.204]
  0-6 hours post-dose | 23.851 (1.057) [lower limit 1.057] | 28.632 (1.053) [lower limit 1.053] | 24.381 (1.058) [lower limit 1.058] | 4.024 (1.812) [lower limit 1.812] | 6.308 (1.849) [lower limit 1.849]
  0-12 hours post-dose | 44.207 (2.266) [lower limit 2.266] | 51.737 (2.258) [lower limit 2.258] | 42.907 (2.268) [lower limit 2.268] | 7.003 (3.883) [lower limit 3.883] | 13.455 (3.964) [lower limit 3.964]
  0-24 hours post-dose | 77.596 (4.949) [lower limit 4.949] | 83.884 (4.930) [lower limit 4.930] | 72.796 (4.953) [lower limit 4.953] | 12.533 (8.481) [lower limit 8.481] | 28.400 (8.656) [lower limit 8.656]
Statistical Analysis 1: Comparison: Naproxen Sodium/ Caffeine 220/65 mg vs Naproxen Sodium/Caffeine 2x220/65 mg; 0-2 hours post-dose; Test type: Other; p < 0.001, ANCOVA; Geometric LS means = -1.602, 95% CI 2-sided [-2.548 to -0.656]
Statistical Analysis 2: Comparison: Naproxen Sodium/Caffeine 2x220/65 mg vs Naproxen Sodium 220 mg; 0-2 hours post-dose; Test type: Other; p = 0.043, ANCOVA; Geometric LS means = 0.976, 95% CI 2-sided [0.029 to 1.923]
Statistical Analysis 3: Comparison: Naproxen Sodium 220 mg vs Caffeine 100 mg; 0-2 hours post-dose; Test type: Other; p < 0.001, ANCOVA; Geometric LS means = 6.097, 95% CI 2-sided [4.766 to 7.427]
Statistical Analysis 4: Comparison: Caffeine 100 mg vs Placebo; 0-2 hours post-dose; Test type: Other; p = 0.711, ANCOVA; Geometric LS means = 0.31, 95% CI 2-sided [-1.332 to 1.951]
Statistical Analysis 5: Comparison: Naproxen Sodium/ Caffeine 220/65 mg vs Naproxen Sodium 220 mg; 0-2 hours post-dose; Test type: Other; p = 0.196, ANCOVA; Geometric LS means = -0.626, 95% CI 2-sided [-1.575 to 0.323]
Statistical Analysis 6: Comparison: Naproxen Sodium/Caffeine 2x220/65 mg vs Caffeine 100 mg; 0-2 hours post-dose; Test type: Other; p < 0.001, ANCOVA; Geometric LS means = 7.073, 95% CI 2-sided [5.744 to 8.402]
Statistical Analysis 7: Comparison: Naproxen Sodium 220 mg vs Placebo; 0-2 hours post-dose; Test type: Other; p < 0.001, ANCOVA; Geometric LS means = 6.406, 95% CI 2-sided [5.055 to 7.757]
Statistical Analysis 8: Comparison: Naproxen Sodium/ Caffeine 220/65 mg vs Caffeine 100 mg; 0-2 hours post-dose; Test type: Other; p < 0.001, ANCOVA; Geometric LS means = 5.471, 95% CI 2-sided [4.141 to 6.801]
Statistical Analysis 9: Comparison: Naproxen Sodium/Caffeine 2x220/65 mg vs Placebo; 0-2 hours post-dose; Test type: Other; p < 0.001, ANCOVA; Geometric LS means = 7.383, 95% CI 2-sided [6.033 to 8.732]
Statistical Analysis 10: Comparison: Naproxen Sodium/ Caffeine 220/65 mg vs Placebo; 0-2 hours post-dose; Test type: Other; p < 0.001, ANCOVA; Geometric LS means = 5.78, 95% CI 2-sided [4.43 to 7.131]

3. Secondary Outcome: Total Pain Relief (TOTPAR) From 0 to 2, 4, 6, 8, 12 and 24 Hours Post-dose
Description: Total Pain Relief (TOTPAR) is a cumulative measure that evaluates the overall pain relief over a specific time frame from 0-2,0-4,0-6,0-8,0-12 and 0-24 following drug administration. It is calculated by multiplying the pain relief score from the categorical pain relief scale at each time post-dose time by multiplying the duration (in hours) since the preceding time point and then adding these values. Categorical Pain Relief Scale measure the degree of pain relief using a scale from 0 to 4, in which 0 is no relief, 1 a little relief, 2 some relief, 3 a lot of relief and 4 complete relief. Higher values of TOTPAR indicates better pain relief and suggest that the investigational product provided consistence and meaningful pain relief over the period. Low TOTPAR values indicates minimal pain relief or short-lasting efficacy.
Time Frame: up to 24 hours post-dose
Measure: Least Squares Mean (Standard Error); unit: Points on scale
Arm/Group | Naproxen Sodium/ Caffeine 220/65 mg | Naproxen Sodium/Caffeine 2x220/65 mg | Naproxen Sodium 220 mg | Caffeine 100 mg | Placebo
Number analyzed (Participants) | 147 | 148 | 147 | 50 | 49
Points on scale
  0-2 hours post-dose | 3.284 (0.114) [lower limit 0.114] | 3.870 (0.114) [lower limit 0.114] | 3.417 (0.115) [lower limit 0.115] | 1.047 (0.196) [lower limit 0.196] | 1.216 (0.200) [lower limit 0.200]
  0-4 hours post-dose | 7.781 (0.287) [lower limit 0.287] | 9.118 (0.286) [lower limit 0.286] | 8.102 (0.287) [lower limit 0.287] | 2.120 (0.492) [lower limit 0.492] | 3.168 (0.502) [lower limit 0.502]
  0-6 hours post-dose | 12.098 (0.465) [lower limit 0.465] | 14.061 (0.464) [lower limit 0.464] | 12.420 (0.466) [lower limit 0.466] | 3.228 (0.798) [lower limit 0.798] | 4.870 (0.814) [lower limit 0.814]
  0-8 hours post-dose | 16.227 (0.645) [lower limit 0.645] | 18.625 (0.642) [lower limit 0.642] | 16.225 (0.645) [lower limit 0.645] | 4.327 (1.105) [lower limit 1.105] | 6.552 (1.128) [lower limit 1.128]
  0-12 hours post-dose | 23.512 (1.029) [lower limit 1.029] | 26.461 (1.026) [lower limit 1.026] | 22.767 (1.030) [lower limit 1.030] | 6.264 (1.764) [lower limit 1.764] | 9.700 (1.801) [lower limit 1.801]
  0-24 hours post-dose | 41.596 (2.281) [lower limit 2.281] | 43.908 (2.272) [lower limit 2.272] | 39.127 (2.283) [lower limit 2.283] | 12.047 (3.909) [lower limit 3.909] | 18.975 (3.990) [lower limit 3.990]
Statistical Analysis 1: Comparison: Naproxen Sodium/ Caffeine 220/65 mg vs Naproxen Sodium/Caffeine 2x220/65 mg; 0-2 hours post-dose; Test type: Other; p < 0.001, ANCOVA; Geometric LS means = -0.586, 95% CI 2-sided [-0.903 to -0.269]
Statistical Analysis 2: Comparison: Naproxen Sodium/Caffeine 2x220/65 mg vs Naproxen Sodium 220 mg; 0-2 hours post-dose; Test type: Other; p = 0.005, ANCOVA; Geometric LS means = 0.454, 95% CI 2-sided [0.136 to 0.771]
Statistical Analysis 3: Comparison: Naproxen Sodium 220 mg vs Caffeine 100 mg; 0-2 hours post-dose; Test type: Other; p < 0.001, ANCOVA; Geometric LS means = 2.369, 95% CI 2-sided [1.923 to 2.815]
Statistical Analysis 4: Comparison: Caffeine 100 mg vs Placebo; 0-2 hours post-dose; Test type: Other; p = 0.548, ANCOVA; Geometric LS means = -0.169, 95% CI 2-sided [-0.719 to 0.382]
Statistical Analysis 5: Comparison: Naproxen Sodium/ Caffeine 220/65 mg vs Naproxen Sodium 220 mg; 0-2 hours post-dose; Test type: Other; p = 0.415, ANCOVA; Geometric LS means = -0.132, 95% CI 2-sided [-0.451 to 0.186]
Statistical Analysis 6: Comparison: Naproxen Sodium/Caffeine 2x220/65 mg vs Caffeine 100 mg; 0-2 hours post-dose; Test type: Other; p < 0.001, ANCOVA; Geometric LS means = 2.823, 95% CI 2-sided [2.377 to 3.268]
Statistical Analysis 7: Comparison: Naproxen Sodium 220 mg vs Placebo; 0-2 hours post-dose; Test type: Other; p < 0.001, ANCOVA; Geometric LS means = 2.201, 95% CI 2-sided [1.748 to 2.654]
Statistical Analysis 8: Comparison: Naproxen Sodium/ Caffeine 220/65 mg vs Caffeine 100 mg; 0-2 hours post-dose; Test type: Other; p < 0.001, ANCOVA; Geometric LS means = 2.237, 95% CI 2-sided [1.791 to 2.683]
Statistical Analysis 9: Comparison: Naproxen Sodium/Caffeine 2x220/65 mg vs Placebo; 0-2 hours post-dose; Test type: Other; p < 0.001, ANCOVA; Geometric LS means = 2.654, 95% CI 2-sided [2.202 to 3.106]
Statistical Analysis 10: Comparison: Naproxen Sodium/Caffeine 2x220/65 mg vs Placebo; 0-2 hours post-dose; Test type: Other; p < 0.001, ANCOVA; Geometric LS means = 2.068, 95% CI 2-sided [1.615 to 2.521]
Statistical Analysis 11: Comparison: Naproxen Sodium/ Caffeine 220/65 mg vs Naproxen Sodium/Caffeine 2x220/65 mg; 0-4 hours post-dose; Test type: Other; p < 0.001, ANCOVA; Geometric LS means = -1.338, 95% CI 2-sided [-2.133 to -0.542]
Statistical Analysis 12: Comparison: Naproxen Sodium/Caffeine 2x220/65 mg vs Naproxen Sodium 220 mg; 0-4 hours post-dose; Test type: Other; p = 0.012, ANCOVA; Geometric LS means = 1.016, 95% CI 2-sided [0.22 to 1.813]
Statistical Analysis 13: Comparison: Naproxen Sodium 220 mg vs Caffeine 100 mg; 0-4 hours post-dose; Test type: Other; p < 0.001, ANCOVA; Geometric LS means = 5.982, 95% CI 2-sided [4.864 to 7.101]
Statistical Analysis 14: Comparison: Caffeine 100 mg vs Placebo; 0-4 hours post-dose; Test type: Other; p = 0.136, ANCOVA; Geometric LS means = -1.048, 95% CI 2-sided [-2.428 to 0.332]
Statistical Analysis 15: Comparison: Naproxen Sodium/ Caffeine 220/65 mg vs Naproxen Sodium 220 mg; 0-4 hours post-dose; Test type: Other; p = 0.43, ANCOVA; Geometric LS means = -0.321, 95% CI 2-sided [-1.119 to 0.477]
Statistical Analysis 16: Comparison: Naproxen Sodium/Caffeine 2x220/65 mg vs Caffeine 100 mg; 0-4 hours post-dose; Test type: Other; p < 0.001, ANCOVA; Geometric LS means = 6.999, 95% CI 2-sided [5.881 to 8.116]
Statistical Analysis 17: Comparison: Naproxen Sodium 220 mg vs Placebo; 0-4 hours post-dose; Test type: Other; p < 0.001, ANCOVA; Geometric LS means = 4.934, 95% CI 2-sided [3.798 to 6.07]
Statistical Analysis 18: Comparison: Naproxen Sodium/ Caffeine 220/65 mg vs Caffeine 100 mg; 0-4 hours post-dose; Test type: Other; p < 0.001, ANCOVA; Geometric LS means = 5.661, 95% CI 2-sided [4.543 to 6.779]
Statistical Analysis 19: Comparison: Naproxen Sodium/Caffeine 2x220/65 mg vs Placebo; 0-4 hours post-dose; Test type: Other; p < 0.001, ANCOVA; Geometric LS means = 5.951, 95% CI 2-sided [4.816 to 7.085]
Statistical Analysis 20: Comparison: Naproxen Sodium/ Caffeine 220/65 mg vs Placebo; 0-4 hours post-dose; Test type: Other; p < 0.001, ANCOVA; Geometric LS means = 4.613, 95% CI 2-sided [3.478 to 5.749]
Statistical Analysis 21: Comparison: Naproxen Sodium/ Caffeine 220/65 mg vs Naproxen Sodium/Caffeine 2x220/65 mg; 0-6 hours post-dose; Test type: Other; p = 0.003, ANCOVA; Geometric LS means = -1.963, 95% CI 2-sided [-3.254 to -0.673]
Statistical Analysis 22: Comparison: Naproxen Sodium/Caffeine 2x220/65 mg vs Naproxen Sodium 220 mg; 0-6 hours post-dose; Test type: Other; p = 0.013, ANCOVA; Geometric LS means = 1.641, 95% CI 2-sided [0.35 to 2.933]
Statistical Analysis 23: Comparison: Naproxen Sodium 220 mg vs Caffeine 100 mg; 0-6 hours post-dose; Test type: Other; p < 0.001, ANCOVA; Geometric LS means = 9.191, 95% CI 2-sided [7.377 to 11.006]
Statistical Analysis 24: Comparison: Caffeine 100 mg vs Placebo; 0-6 hours post-dose; Test type: Other; p = 0.15, ANCOVA; Geometric LS means = -1.642, 95% CI 2-sided [-3.881 to 0.597]
Statistical Analysis 25: Comparison: Naproxen Sodium/ Caffeine 220/65 mg vs Naproxen Sodium 220 mg; 0-6 hours post-dose; Test type: Other; p = 0.625, ANCOVA; Geometric LS means = -0.322, 95% CI 2-sided [-1.617 to 0.972]
Statistical Analysis 26: Comparison: Naproxen Sodium/Caffeine 2x220/65 mg vs Caffeine 100 mg; 0-6 hours post-dose; Test type: Other; p < 0.001, ANCOVA; Geometric LS means = 10.833, 95% CI 2-sided [9.02 to 12.645]
Statistical Analysis 27: Comparison: Naproxen Sodium 220 mg vs Placebo; 0-6 hours post-dose; Test type: Other; p < 0.001, ANCOVA; Geometric LS means = 7.55, 95% CI 2-sided [5.707 to 9.392]
Statistical Analysis 28: Comparison: Naproxen Sodium/ Caffeine 220/65 mg vs Caffeine 100 mg; 0-6 hours post-dose; Test type: Other; p < 0.001, ANCOVA; Geometric LS means = 8.869, 95% CI 2-sided [7.055 to 10.683]
Statistical Analysis 29: Comparison: Naproxen Sodium/Caffeine 2x220/65 mg vs Placebo; 0-6 hours post-dose; Test type: Other; p < 0.001, ANCOVA; Geometric LS means = 9.191, 95% CI 2-sided [7.351 to 11.031]
Statistical Analysis 30: Comparison: Naproxen Sodium/ Caffeine 220/65 mg vs Placebo; 0-6 hours post-dose; Test type: Other; p < 0.001, ANCOVA; Geometric LS means = 7.228, 95% CI 2-sided [5.386 to 9.07]
Statistical Analysis 31: Comparison: Naproxen Sodium/ Caffeine 220/65 mg vs Naproxen Sodium/Caffeine 2x220/65 mg; 0-8 hours post-dose; Test type: Other; p = 0.009, ANCOVA; Geometric LS means = -2.398, 95% CI 2-sided [-4.185 to -0.61]
Statistical Analysis 32: Comparison: Naproxen Sodium/Caffeine 2x220/65 mg vs Naproxen Sodium 220 mg; 0-8 hours post-dose; Test type: Other; p = 0.009, ANCOVA; Geometric LS means = 2.4, 95% CI 2-sided [0.61 to 4.189]
Statistical Analysis 33: Comparison: Naproxen Sodium 220 mg vs Caffeine 100 mg; 0-8 hours post-dose; Test type: Other; p < 0.001, ANCOVA; Geometric LS means = 11.898, 95% CI 2-sided [9.384 to 14.412]
Statistical Analysis 34: Comparison: Caffeine 100 mg vs Placebo; 0-8 hours post-dose; Test type: Other; p = 0.159, ANCOVA; Geometric LS means = -2.225, 95% CI 2-sided [-5.327 to 0.877]
Statistical Analysis 35: Comparison: Naproxen Sodium/ Caffeine 220/65 mg vs Naproxen Sodium 220 mg; 0-8 hours post-dose; Test type: Other; p = 0.998, ANCOVA; Geometric LS means = 0.002, 95% CI 2-sided [-1.792 to 1.795]
Statistical Analysis 36: Comparison: Naproxen Sodium/Caffeine 2x220/65 mg vs Caffeine 100 mg; 0-8 hours post-dose; Test type: Other; p < 0.001, ANCOVA; Geometric LS means = 14.298, 95% CI 2-sided [11.787 to 16.809]
Statistical Analysis 37: Comparison: Naproxen Sodium 220 mg vs Placebo; 0-8 hours post-dose; Test type: Other; p < 0.001, ANCOVA; Geometric LS means = 9.673, 95% CI 2-sided [7.12 to 12.226]
Statistical Analysis 38: Comparison: Naproxen Sodium/ Caffeine 220/65 mg vs Caffeine 100 mg; 0-8 hours post-dose; Test type: Other; p < 0.001, ANCOVA; Geometric LS means = 11.9, 95% CI 2-sided [9.387 to 14.413]
Statistical Analysis 39: Comparison: Naproxen Sodium/Caffeine 2x220/65 mg vs Placebo; 0-8 hours post-dose; Test type: Other; p < 0.001, ANCOVA; Geometric LS means = 12.073, 95% CI 2-sided [9.523 to 14.623]
Statistical Analysis 40: Comparison: Naproxen Sodium/ Caffeine 220/65 mg vs Placebo; 0-8 hours post-dose; Test type: Other; p < 0.001, ANCOVA; Geometric LS means = 9.675, 95% CI 2-sided [7.123 to 12.227]
Statistical Analysis 41: Comparison: Naproxen Sodium/ Caffeine 220/65 mg vs Naproxen Sodium/Caffeine 2x220/65 mg; 0-12 hours post-dose; Test type: Other; p = 0.043, ANCOVA; Geometric LS means = -2.949, 95% CI 2-sided [-5.803 to -0.095]
Statistical Analysis 42: Comparison: Naproxen Sodium/Caffeine 2x220/65 mg vs Naproxen Sodium 220 mg; 0-12 hours post-dose; Test type: Other; p = 0.011, ANCOVA; Geometric LS means = 3.694, 95% CI 2-sided [0.837 to 6.55]
Statistical Analysis 43: Comparison: Naproxen Sodium 220 mg vs Caffeine 100 mg; 0-12 hours post-dose; Test type: Other; p < 0.001, ANCOVA; Geometric LS means = 16.504, 95% CI 2-sided [12.49 to 20.517]
Statistical Analysis 44: Comparison: Caffeine 100 mg vs Placebo; 0-12 hours post-dose; Test type: Other; p = 0.173, ANCOVA; Geometric LS means = -3.437, 95% CI 2-sided [-8.389 to 1.515]
Statistical Analysis 45: Comparison: Naproxen Sodium/ Caffeine 220/65 mg vs Naproxen Sodium 220 mg; 0-12 hours post-dose; Test type: Other; p = 0.61, ANCOVA; Geometric LS means = 0.744, 95% CI 2-sided [-2.119 to 3.608]
Statistical Analysis 46: Comparison: Naproxen Sodium/Caffeine 2x220/65 mg vs Caffeine 100 mg; 0-12 hours post-dose; Test type: Other; p < 0.001, ANCOVA; Geometric LS means = 20.197, 95% CI 2-sided [16.189 to 24.206]
Statistical Analysis 47: Comparison: Naproxen Sodium 220 mg vs Placebo; 0-12 hours post-dose; Test type: Other; p < 0.001, ANCOVA; Geometric LS means = 13.067, 95% CI 2-sided [8.992 to 17.143]
Statistical Analysis 48: Comparison: Naproxen Sodium/Caffeine 2x220/65 mg vs Caffeine 100 mg; 0-12 hours post-dose; Test type: Other; p < 0.001, ANCOVA; Geometric LS means = 17.248, 95% CI 2-sided [13.236 to 21.261]
Statistical Analysis 49: Comparison: Naproxen Sodium/Caffeine 2x220/65 mg vs Placebo; 0-12 hours post-dose; Test type: Other; p < 0.001, ANCOVA; Geometric LS means = 16.761, 95% CI 2-sided [12.69 to 20.831]
Statistical Analysis 50: Comparison: Naproxen Sodium/ Caffeine 220/65 mg vs Placebo; 0-12 hours post-dose; Test type: Other; p < 0.001, ANCOVA; Geometric LS means = 13.812, 95% CI 2-sided [9.738 to 17.886]
Statistical Analysis 51: Comparison: Naproxen Sodium/ Caffeine 220/65 mg vs Naproxen Sodium/Caffeine 2x220/65 mg; 0-24 hours post-dose; Test type: Other; p = 0.473, ANCOVA; Geometric LS means = -2.312, 95% CI 2-sided [-8.635 to 4.011]
Statistical Analysis 52: Comparison: Naproxen Sodium 220 mg vs Caffeine 100 mg; 0-24 hours post-dose; Test type: Other; p < 0.001, ANCOVA; Geometric LS means = 27.08, 95% CI 2-sided [18.188 to 35.973]
Statistical Analysis 53: Comparison: Caffeine 100 mg vs Placebo; 0-24 hours post-dose; Test type: Other; p = 0.215, ANCOVA; Geometric LS means = -6.928, 95% CI 2-sided [-17.9 to 4.044]
Statistical Analysis 54: Comparison: Naproxen Sodium/ Caffeine 220/65 mg vs Naproxen Sodium 220 mg; 0-24 hours post-dose; Test type: Other; p = 0.445, ANCOVA; Geometric LS means = 2.468, 95% CI 2-sided [-3.876 to 8.813]
Statistical Analysis 55: Comparison: Naproxen Sodium 220 mg vs Placebo; 0-24 hours post-dose; Test type: Other; p < 0.001, ANCOVA; Geometric LS means = 20.152, 95% CI 2-sided [11.122 to 29.183]
Statistical Analysis 56: Comparison: Naproxen Sodium/Caffeine 2x220/65 mg vs Placebo; 0-24 hours post-dose; Test type: Other; p < 0.001, ANCOVA; Geometric LS means = 24.933, 95% CI 2-sided [15.914 to 33.952]
Statistical Analysis 57: Comparison: Naproxen Sodium/ Caffeine 220/65 mg vs Placebo; 0-24 hours post-dose; Test type: Other; p < 0.001, ANCOVA; Geometric LS means = 22.621, 95% CI 2-sided [13.594 to 31.648]

4. Secondary Outcome: Time to First Use of Rescue Medication
Time Frame: Up to 24 hours post-dose
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Naproxen Sodium/ Caffeine 220/65 mg | Naproxen Sodium/Caffeine 2x220/65 mg | Naproxen Sodium 220 mg | Caffeine 100 mg | Placebo
Number analyzed (Participants) | 147 | 148 | 147 | 50 | 49
Hours | NA [17.33 to NA] — Insufficient number of participants with events. | NA [14.08 to NA] — Insufficient number of participants with events. | 19.72 [11.08 to NA] — Insufficient number of participants with events. | 2.07 [1.72 to 2.75] | 2.65 [1.67 to 7.28]
Statistical Analysis 1: Comparison: Naproxen Sodium/ Caffeine 220/65 mg vs Naproxen Sodium/Caffeine 2x220/65 mg; Test type: Other; p = 0.963, ANCOVA
Statistical Analysis 2: Comparison: Naproxen Sodium/Caffeine 2x220/65 mg vs Naproxen Sodium 220 mg; Test type: Other; p = 0.118, ANCOVA
Statistical Analysis 3: Comparison: Naproxen Sodium 220 mg vs Caffeine 100 mg; Test type: Other; p < 0.001, ANCOVA
Statistical Analysis 4: Comparison: Caffeine 100 mg vs Placebo; Test type: Other; p = 0.244, ANCOVA
Statistical Analysis 5: Comparison: Naproxen Sodium/ Caffeine 220/65 mg vs Naproxen Sodium 220 mg; Test type: Other; p = 0.139, ANCOVA
Statistical Analysis 6: Comparison: Naproxen Sodium/ Caffeine 220/65 mg vs Naproxen Sodium 220 mg; Test type: Other; p < 0.001, ANCOVA
Statistical Analysis 7: Comparison: Naproxen Sodium 220 mg vs Placebo; Test type: Other; p < 0.001, ANCOVA
Statistical Analysis 8: Comparison: Naproxen Sodium/ Caffeine 220/65 mg vs Caffeine 100 mg; Test type: Other; p < 0.001, ANCOVA
Statistical Analysis 9: Comparison: Naproxen Sodium/Caffeine 2x220/65 mg vs Placebo; Test type: Other; p < 0.001, ANCOVA
Statistical Analysis 10: Comparison: Naproxen Sodium/ Caffeine 220/65 mg vs Placebo; Test type: Other; p < 0.001, ANCOVA

5. Secondary Outcome: The Cumulative Proportion of Participants Taking Rescue Medication Over the 24 Hour Period
Time Frame: Up to 24 hours post-dose
Measure: Number; unit: proportion
Arm/Group | Naproxen Sodium/ Caffeine 220/65 mg | Naproxen Sodium/Caffeine 2x220/65 mg | Naproxen Sodium 220 mg | Caffeine 100 mg | Placebo
Number analyzed (Participants) | 147 | 148 | 147 | 50 | 49
proportion
  0.5 hour | 0 | 0 | 0 | 0 | 0
  less or equal 1 hour | 0.007 | 0 | 0.007 | 0.04 | 0.02
  less or equal 1.5 hour | 0.027 | 0.007 | 0.007 | 0.3 | 0.2
  less or equal 2 hours | 0.1 | 0.034 | 0.048 | 0.4 | 0.5
  less or equal 3 hours | 0.1 | 0.1 | 0.1 | 0.7 | 0.5
  less or equal 4hours | 0.2 | 0.1 | 0.1 | 0.7 | 0.6
  less or equal 5 hours | 0.2 | 0.1 | 0.1 | 0.7 | 0.6
  less or equal 6 hours | 0.2 | 0.1 | 0.2 | 0.8 | 0.6
  less or equal 7 hours | 0.2 | 0.1 | 0.2 | 0.8 | 0.6
  less or equal 8 hours | 0.2 | 0.1 | 0.3 | 0.8 | 0.6
  less or equal 9 hours | 0.3 | 0.2 | 0.3 | 0.8 | 0.7
  less or equal 10 hours | 0.3 | 0.2 | 0.4 | 0.8 | 0.7
  less or equal 11 hours | 0.4 | 0.3 | 0.4 | 0.8 | 0.7
  less or equal 12 hours | 0.4 | 0.3 | 0.4 | 0.8 | 0.7
  less or equal 14 hours | 0.4 | 0.4 | 0.4 | 0.8 | 0.7
  less or equal 16 hours | 0.4 | 0.4 | 0.5 | 0.8 | 0.7
  less or equal 18 hours | 0.4 | 0.4 | 0.5 | 0.8 | 0.7
  less or equal 20 hours | 0.4 | 0.4 | 0.5 | 0.8 | 0.7
  less or equal 22 hours | 0.4 | 0.4 | 0.5 | 0.8 | 0.7
  less or equal 24 hours | 0.4 | 0.4 | 0.5 | 0.8 | 0.7

6. Secondary Outcome: Time to First Perceptible Relief Measured by a Stopwatch
Time Frame: Up to 24 hours post-dose
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Naproxen Sodium/ Caffeine 220/65 mg | Naproxen Sodium/Caffeine 2x220/65 mg | Naproxen Sodium 220 mg | Caffeine 100 mg | Placebo
Number analyzed (Participants) | 147 | 148 | 147 | 50 | 49
Hours | 0.39 [0.33 to 0.42] | 0.35 [0.32 to 0.41] | 0.35 [0.32 to 0.39] | 0.60 [0.42 to 4.13] | 1.93 [0.51 to NA] — Insufficient number of participants with events.
Statistical Analysis 1: Comparison: Naproxen Sodium/ Caffeine 220/65 mg vs Naproxen Sodium/Caffeine 2x220/65 mg; Test type: Other; p = 0.647, ANCOVA
Statistical Analysis 2: Comparison: Naproxen Sodium/Caffeine 2x220/65 mg vs Naproxen Sodium 220 mg; Test type: Other; p = 0.714, ANCOVA
Statistical Analysis 3: Comparison: Caffeine 100 mg vs Placebo; Test type: Other; p = 0.065, ANCOVA
Statistical Analysis 4: Comparison: Naproxen Sodium/ Caffeine 220/65 mg vs Naproxen Sodium 220 mg; Test type: Other; p = 0.742, ANCOVA
Statistical Analysis 5: Comparison: Naproxen Sodium/Caffeine 2x220/65 mg vs Caffeine 100 mg; Test type: Other; p < 0.001, ANCOVA
Statistical Analysis 6: Comparison: Naproxen Sodium 220 mg vs Placebo; Test type: Other; p < 0.001, ANCOVA
Statistical Analysis 7: Comparison: Naproxen Sodium/ Caffeine 220/65 mg vs Caffeine 100 mg; Test type: Other; p < 0.001, ANCOVA
Statistical Analysis 8: Comparison: Naproxen Sodium/Caffeine 2x220/65 mg vs Placebo; Test type: Other; p < 0.001, ANCOVA
Statistical Analysis 9: Comparison: Naproxen Sodium/ Caffeine 220/65 mg vs Placebo; Test type: Other; p < 0.001, ANCOVA

7. Secondary Outcome: Time to Meaningful Relief Measured by a Stopwatch
Description: meaningful relief is the point when the participant perceives their pain as significant and meaningful to them using the double-stopwatched method that allows to differentiate between the onset of the analgesic effect (first perceptible pain relief) and the onset of meaningful pain relief
Time Frame: Up to 24 hours post-dose
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Naproxen Sodium/ Caffeine 220/65 mg | Naproxen Sodium/Caffeine 2x220/65 mg | Naproxen Sodium 220 mg | Caffeine 100 mg | Placebo
Number analyzed (Participants) | 147 | 148 | 147 | 50 | 49
Hours | 0.83 [0.71 to 0.92] | 0.76 [0.67 to 0.85] | 0.79 [0.67 to 0.93] | NA [2.24 to NA] — Insufficient number of participants with events. | 5.63 [2.11 to 5.78]
Statistical Analysis 1: Comparison: Naproxen Sodium/ Caffeine 220/65 mg vs Naproxen Sodium/Caffeine 2x220/65 mg; Test type: Other; p = 0.162, ANCOVA
Statistical Analysis 2: Comparison: Naproxen Sodium/Caffeine 2x220/65 mg vs Naproxen Sodium 220 mg; Test type: Other; p = 0.319, ANCOVA
Statistical Analysis 3: Comparison: Naproxen Sodium 220 mg vs Caffeine 100 mg; Test type: Other; p < 0.001, ANCOVA
Statistical Analysis 4: Comparison: Caffeine 100 mg vs Placebo; Test type: Other; p = 0.343, ANCOVA
Statistical Analysis 5: Comparison: Naproxen Sodium/Caffeine 2x220/65 mg vs Caffeine 100 mg; Test type: Other; p < 0.001, ANCOVA
Statistical Analysis 6: Comparison: Naproxen Sodium 220 mg vs Placebo; Test type: Other; p < 0.001, ANCOVA
Statistical Analysis 7: Comparison: Naproxen Sodium/ Caffeine 220/65 mg vs Caffeine 100 mg; Test type: Other; p < 0.001, ANCOVA
Statistical Analysis 8: Comparison: Naproxen Sodium/Caffeine 2x220/65 mg vs Placebo; Test type: Other; p < 0.001, ANCOVA
Statistical Analysis 9: Comparison: Naproxen Sodium/ Caffeine 220/65 mg vs Placebo; Test type: Other; p < 0.001, ANCOVA

8. Secondary Outcome: Time to First Perceptible Relief Confirmed by Meaningful Relief Defined as the Time to Perceptible Pain Relief
Time Frame: Up to 24 hours post-dose
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Naproxen Sodium/ Caffeine 220/65 mg | Naproxen Sodium/Caffeine 2x220/65 mg | Naproxen Sodium 220 mg | Caffeine 100 mg | Placebo
Number analyzed (Participants) | 147 | 148 | 147 | 50 | 49
Hours | 0.83 [0.71 to 0.92] | 0.76 [0.67 to 0.85] | 0.79 [0.67 to 0.93] | NA [2.24 to NA] — Insufficient number of participants with events. | 5.63 [2.11 to 5.78]
Statistical Analysis 1: Comparison: Naproxen Sodium/ Caffeine 220/65 mg vs Naproxen Sodium/Caffeine 2x220/65 mg; Test type: Other; p = 0.162, ANCOVA
Statistical Analysis 2: Comparison: Naproxen Sodium/Caffeine 2x220/65 mg vs Naproxen Sodium 220 mg; Test type: Other; p = 0.319, ANCOVA
Statistical Analysis 3: Comparison: Naproxen Sodium 220 mg vs Caffeine 100 mg; Test type: Other; p < 0.001, ANCOVA
Statistical Analysis 4: Comparison: Caffeine 100 mg vs Placebo; Test type: Other; p = 0.343, ANCOVA
Statistical Analysis 5: Comparison: Naproxen Sodium 220 mg vs Placebo; Test type: Other; p = 0.772, ANCOVA
Statistical Analysis 6: Comparison: Naproxen Sodium/Caffeine 2x220/65 mg vs Caffeine 100 mg; Test type: Other; p < 0.001, ANCOVA
Statistical Analysis 7: Comparison: Naproxen Sodium 220 mg vs Placebo; Test type: Other; p < 0.001, ANCOVA
Statistical Analysis 8: Comparison: Naproxen Sodium/ Caffeine 220/65 mg vs Caffeine 100 mg; Test type: Other; p < 0.001, ANCOVA
Statistical Analysis 9: Comparison: Naproxen Sodium/Caffeine 2x220/65 mg vs Placebo; Test type: Other; p < 0.001, ANCOVA
Statistical Analysis 10: Comparison: Naproxen Sodium/ Caffeine 220/65 mg vs Placebo; Test type: Other; p < 0.001, ANCOVA

9. Secondary Outcome: Pain Intensity Difference (PID)
Description: Pain Intensity Difference (PID) is the change of pain intensity at a specific time point compared to baseline using the Numerical Rating Scale from 0 to 10. Value of 0 score means no pain and 10 score result means the worst possible pain. For each post-dose time point, pain intensity differences will be derived by subtracting the pain intensity at the post-dose time point from the baseline intensity score. Positive PID values indicate pain relief (reduction in pain intensity), while negative or small PID values suggest little or no reduction in pain intensity
Time Frame: up to 24 hours post-dose
Measure: Mean (Standard Deviation); unit: Points on scale
Arm/Group | Naproxen Sodium/ Caffeine 220/65 mg | Naproxen Sodium/Caffeine 2x220/65 mg | Naproxen Sodium 220 mg | Caffeine 100 mg | Placebo
Number analyzed (Participants) | 147 | 148 | 147 | 50 | 49
Points on scale
  Baseline | 7.6 (1.22) [lower limit 1.22] | 7.6 (1.20) [lower limit 1.20] | 7.8 (1.21) [lower limit 1.21] | 7.7 (1.39) [lower limit 1.39] | 7.7 (0.99) [lower limit 0.99]
  0.5 hours post-dose | 1.8 (1.89) [lower limit 1.89] | 2.3 (1.91) [lower limit 1.91] | 2.4 (1.98) [lower limit 1.98] | 1.0 (1.38) [lower limit 1.38] | 0.6 (1.18) [lower limit 1.18]
  1 hour post-dose | 3.4 (2.40) [lower limit 2.40] | 4.3 (2.18) [lower limit 2.18] | 3.7 (2.23) [lower limit 2.23] | 0.8 (1.67) [lower limit 1.67] | 0.7 (1.89) [lower limit 1.89]
  1.5 hours post-dose | 4.0 (2.40) [lower limit 2.40] | 4.9 (2.13) [lower limit 2.13] | 4.3 (2.27) [lower limit 2.27] | 0.6 (1.68) [lower limit 1.68] | 0.6 (2.17) [lower limit 2.17]
  2 hours post-dose | 4.4 (2.56) [lower limit 2.56] | 5.2 (2.12) [lower limit 2.12] | 4.7 (2.30) [lower limit 2.30] | 0.7 (1.99) [lower limit 1.99] | 0.9 (2.48) [lower limit 2.48]
  3 hours post-dose | 4.3 (2.55) [lower limit 2.55] | 5.2 (2.28) [lower limit 2.28] | 4.4 (2.45) [lower limit 2.45] | 0.4 (1.94) [lower limit 1.94] | 1.1 (2.64) [lower limit 2.64]
  4 hours post-dose | 4.2 (2.54) [lower limit 2.54] | 5.1 (2.47) [lower limit 2.47] | 4.3 (2.65) [lower limit 2.65] | 0.6 (2.19) [lower limit 2.19] | 1.4 (2.99) [lower limit 2.99]
  5 hours post-dose | 4.0 (2.55) [lower limit 2.55] | 4.8 (2.46) [lower limit 2.46] | 4.1 (2.73) [lower limit 2.73] | 0.5 (2.11) [lower limit 2.11] | 1.2 (2.84) [lower limit 2.84]
  6 hours post-dose | 3.9 (2.60) [lower limit 2.60] | 4.6 (2.48) [lower limit 2.48] | 3.8 (2.74) [lower limit 2.74] | 0.6 (2.34) [lower limit 2.34] | 1.2 (3.01) [lower limit 3.01]
  7 hours post-dose | 3.8 (2.61) [lower limit 2.61] | 4.4 (2.56) [lower limit 2.56] | 3.5 (2.80) [lower limit 2.80] | 0.6 (2.30) [lower limit 2.30] | 1.2 (2.94) [lower limit 2.94]
  8 hours post-dose | 3.6 (2.63) [lower limit 2.63] | 4.1 (2.60) [lower limit 2.60] | 3.3 (2.88) [lower limit 2.88] | 0.6 (2.30) [lower limit 2.30] | 1.2 (3.00) [lower limit 3.00]
  9 hours post dose | 3.5 (2.72) [lower limit 2.72] | 3.9 (2.68) [lower limit 2.68] | 3.3 (2.96) [lower limit 2.96] | 0.6 (2.47) [lower limit 2.47] | 1.3 (3.15) [lower limit 3.15]
  10 hours post-dose | 3.3 (2.78) [lower limit 2.78] | 3.8 (2.81) [lower limit 2.81] | 3.1 (3.03) [lower limit 3.03] | 0.4 (2.25) [lower limit 2.25] | 1.3 (3.24) [lower limit 3.24]
  11 hours post-dose | 3.1 (2.84) [lower limit 2.84] | 3.6 (2.86) [lower limit 2.86] | 2.9 (3.02) [lower limit 3.02] | 0.4 (2.34) [lower limit 2.34] | 1.2 (3.23) [lower limit 3.23]
  12 hours post-dose | 2.9 (2.90) [lower limit 2.90] | 3.2 (2.90) [lower limit 2.90] | 2.8 (3.07) [lower limit 3.07] | 0.4 (2.29) [lower limit 2.29] | 1.3 (3.32) [lower limit 3.32]
  14 hours post-dose | 2.9 (2.97) [lower limit 2.97] | 2.9 (3.01) [lower limit 3.01] | 2.6 (3.04) [lower limit 3.04] | 0.4 (2.20) [lower limit 2.20] | 1.3 (3.32) [lower limit 3.32]
  16 hours post-dose | 2.6 (2.99) [lower limit 2.99] | 2.7 (2.85) [lower limit 2.85] | 2.4 (3.04) [lower limit 3.04] | 0.4 (2.27) [lower limit 2.27] | 1.2 (3.21) [lower limit 3.21]
  18 hours post-dose | 2.7 (3.05) [lower limit 3.05] | 2.6 (2.83) [lower limit 2.83] | 2.4 (3.02) [lower limit 3.02] | 0.4 (2.27) [lower limit 2.27] | 1.2 (3.22) [lower limit 3.22]
  20 hours post-dose | 2.7 (3.07) [lower limit 3.07] | 2.6 (2.81) [lower limit 2.81] | 2.5 (3.06) [lower limit 3.06] | 0.4 (2.33) [lower limit 2.33] | 1.2 (3.28) [lower limit 3.28]
  22 hours post-dose | 2.8 (3.19) [lower limit 3.19] | 2.7 (2.85) [lower limit 2.85] | 2.6 (3.14) [lower limit 3.14] | 0.5 (2.55) [lower limit 2.55] | 1.4 (3.51) [lower limit 3.51]
  24 hours post-dose | 2.9 (3.19) [lower limit 3.19] | 2.8 (2.92) [lower limit 2.92] | 2.6 (3.20) [lower limit 3.20] | 0.6 (2.62) [lower limit 2.62] | 1.5 (3.63) [lower limit 3.63]

10. Secondary Outcome: Pain Relief Score
Description: Pain Relief Score (PRS): 0 = No Relief; 1 = A Little Relief; 2 = Some Relief; 3 = A Lot of Relief; 4 = Complete Relief.
Time Frame: Up to 24 hours post-dose
Measure: Mean (Standard Deviation); unit: Points on scale
Arm/Group | Naproxen Sodium/ Caffeine 220/65 mg | Naproxen Sodium/Caffeine 2x220/65 mg | Naproxen Sodium 220 mg | Caffeine 100 mg | Placebo
Number analyzed (Participants) | 147 | 148 | 147 | 50 | 49
Points on scale
  0.5 hours post-dose | 1.3 (0.93) [lower limit 0.93] | 1.5 (1.01) [lower limit 1.01] | 1.5 (0.97) [lower limit 0.97] | 0.7 (0.72) [lower limit 0.72] | 0 (0.65) [lower limit 0.65]
  1 hour post-dose | 2.0 (1.04) [lower limit 1.04] | 2.4 (0.9) [lower limit 0.9] | 2.1 (0.99) [lower limit 0.99] | 0.7 (0.9) [lower limit 0.9] | 0.8 (0.96) [lower limit 0.96]
  1.5 hours post-dose | 2.3 (1.07) [lower limit 1.07] | 2.6 (0.87) [lower limit 0.87] | 2.3 (0.94) [lower limit 0.94] | 0.6 (0.88) [lower limit 0.88] | 0.8 (1.04) [lower limit 1.04]
  2 hours post-dose | 2.3 (1.13) [lower limit 1.13] | 2.7 (0.93) [lower limit 0.93] | 2.5 (0.99) [lower limit 0.99] | 0.7 (0.95) [lower limit 0.95] | 0.9 (1.17) [lower limit 1.17]
  3 hours post-dose | 2.3 (1.19) [lower limit 1.19] | 2.7 (1.06) [lower limit 1.06] | 2.4 (1.11) [lower limit 1.11] | 0.5 (0.93) [lower limit 0.93] | 1.0 (1.25) [lower limit 1.25]
  4 hours post-dose | 2.2 (1.2) [lower limit 1.2] | 2.6 (1.18) [lower limit 1.18] | 2.3 (1.2) [lower limit 1.2] | 0.6 (0.99) [lower limit 0.99] | 1.0 (1.35) [lower limit 1.35]
  5 hours post-dose | 2.1 (1.24) [lower limit 1.24] | 2.5 (1.13) [lower limit 1.13] | 2.3 (1.28) [lower limit 1.28] | 0.5 (1.03) [lower limit 1.03] | 0.8 (1.17) [lower limit 1.17]
  6 hours post-dose | 2.2 (1.26) [lower limit 1.26] | 2.5 (1.12) [lower limit 1.12] | 2.1 (1.28) [lower limit 1.28] | 0.6 (1.07) [lower limit 1.07] | 0.9 (1.3) [lower limit 1.3]
  7 hours post-dose | 2.1 (1.27) [lower limit 1.27] | 2.3 (1.16) [lower limit 1.16] | 2.0 (1.28) [lower limit 1.28] | 0.6 (1.07) [lower limit 1.07] | 0.9 (1.28) [lower limit 1.28]
  8 hours post-dose | 2.1 (1.28) [lower limit 1.28] | 2.2 (1.23) [lower limit 1.23] | 1.8 (1.36) [lower limit 1.36] | 0.5 (1.03) [lower limit 1.03] | 0.8 (1.21) [lower limit 1.21]
  9 hours post-dose | 2.0 (1.33) [lower limit 1.33] | 2.1 (1.28) [lower limit 1.28] | 1.8 (1.39) [lower limit 1.39] | 0.5 (1.02) [lower limit 1.02] | 0.8 (1.28) [lower limit 1.28]
  10 hours post-dose | 1.9 (1.35) [lower limit 1.35] | 2.1 (1.35) [lower limit 1.35] | 1.7 (1.42) [lower limit 1.42] | 0.5 (1.05) [lower limit 1.05] | 0.8 (1.31) [lower limit 1.31]
  11 hours post-dose | 1.8 (1.38) [lower limit 1.38] | 2.0 (1.41) [lower limit 1.41] | 1.6 (1.45) [lower limit 1.45] | 0.5 (1.07) [lower limit 1.07] | 0.8 (1.34) [lower limit 1.34]
  12 hours post-dose | 1.7 (1.4) [lower limit 1.4] | 1.8 (1.46) [lower limit 1.46] | 1.5 (1.47) [lower limit 1.47] | 0.5 (1.07) [lower limit 1.07] | 0.8 (1.34) [lower limit 1.34]
  14 hours post-dose | 1.6 (1.44) [lower limit 1.44] | 1.6 (1.51) [lower limit 1.51] | 1.4 (1.46) [lower limit 1.46] | 0.5 (1.03) [lower limit 1.03] | 0.8 (1.29) [lower limit 1.29]
  16 hours post-dose | 1.5 (1.45) [lower limit 1.45] | 1.5 (1.46) [lower limit 1.46] | 1.3 (1.44) [lower limit 1.44] | 0.5 (1.03) [lower limit 1.03] | 0.7 (1.25) [lower limit 1.25]
  18 hours post-dose | 1.5 (1.45) [lower limit 1.45] | 1.4 (1.44) [lower limit 1.44] | 1.3 (1.43) [lower limit 1.43] | 0.5 (1.03) [lower limit 1.03] | 0.7 (1.25) [lower limit 1.25]
  20 hours post-dose | 1.5 (1.44) [lower limit 1.44] | 1.4 (1.44) [lower limit 1.44] | 1.3 (1.46) [lower limit 1.46] | 0.5 (1.03) [lower limit 1.03] | 0.8 (1.31) [lower limit 1.31]
  22 hours post-dose | 1.5 (1.51) [lower limit 1.51] | 1.5 (1.50) [lower limit 1.50] | 1.4 (1.51) [lower limit 1.51] | 0.5 (1.18) [lower limit 1.18] | 0.9 (1.46) [lower limit 1.46]
  24 hours post-dose | 1.6 (1.53) [lower limit 1.53] | 1.6 (1.51) [lower limit 1.51] | 1.4 (1.56) [lower limit 1.56] | 0.5 (1.22) [lower limit 1.22] | 0.9 (1.51) [lower limit 1.51]

11. Secondary Outcome: Peak Pain Intensity Difference (PID)
Description: The Peak Pain Intensity (peak PID) refers to the maximum change in pain intensity from baseline observed at any post-dose time point using the Numerical Rating Scale from 0 to 10. Value of 0 score means no pain and 10 score result means the worst possible pain. Participants record their pain intensity assessment in the time frame points and the highest value is identified as the Peak Pain Intensity. A high peak pain intensuty (higher value on NRS) indicates severe pain and a less effective analgesic response, and a lower value signifies better pain control and a more effective response.
Time Frame: Up to 24 hours post-dose
Measure: Least Squares Mean (Standard Error); unit: Points on scale
Arm/Group | Naproxen Sodium/ Caffeine 220/65 mg | Naproxen Sodium/Caffeine 2x220/65 mg | Naproxen Sodium 220 mg | Caffeine 100 mg | Placebo
Number analyzed (Participants) | 147 | 148 | 147 | 50 | 49
Points on scale | 6.12 (0.11) [lower limit 0.11] | 6.26 (0.11) [lower limit 0.11] | 6.22 (0.11) [lower limit 0.11] | 6.30 (0.18) [lower limit 0.18] | 6.33 (0.19) [lower limit 0.19]
Statistical Analysis 1: Comparison: Naproxen Sodium/ Caffeine 220/65 mg vs Naproxen Sodium/Caffeine 2x220/65 mg; Test type: Other; p = 0.334, ANCOVA; geometric LS mean square = -0.14, 95% CI 2-sided [-0.44 to 0.15]
Statistical Analysis 2: Comparison: Naproxen Sodium/Caffeine 2x220/65 mg vs Naproxen Sodium 220 mg; Test type: Other; p = 0.783, ANCOVA; geometric LS mean square = 0.04, 95% CI 2-sided [-0.25 to 0.33]
Statistical Analysis 3: Comparison: Naproxen Sodium 220 mg vs Caffeine 100 mg; Test type: Other; p = 0.687, ANCOVA; geometric LS mean square = -0.08, 95% CI 2-sided [-0.5 to 0.33]
Statistical Analysis 4: Comparison: Caffeine 100 mg vs Placebo; Test type: Other; p = 0.927, ANCOVA; geometric LS mean square = -0.02, 95% CI 2-sided [-0.53 to 0.49]
Statistical Analysis 5: Comparison: Naproxen Sodium/ Caffeine 220/65 mg vs Naproxen Sodium 220 mg; Test type: Other; p = 0.492, ANCOVA; geometric LS mean square = -0.1, 95% CI 2-sided [-0.4 to 0.19]
Statistical Analysis 6: Comparison: Naproxen Sodium/Caffeine 2x220/65 mg vs Caffeine 100 mg; Test type: Other; p = 0.836, ANCOVA; geometric LS mean square = -0.04, 95% CI 2-sided [-0.46 to 0.37]
Statistical Analysis 7: Comparison: Naproxen Sodium/ Caffeine 220/65 mg vs Placebo; Test type: Other; p = 0.611, ANCOVA; geometric LS mean square = -0.11, 95% CI 2-sided [-0.53 to 0.31]
Statistical Analysis 8: Comparison: Naproxen Sodium/ Caffeine 220/65 mg vs Caffeine 100 mg; Test type: Other; p = 0.371, ANCOVA; geometric LS mean square = -0.19, 95% CI 2-sided [-0.6 to 0.22]
Statistical Analysis 9: Comparison: Naproxen Sodium/Caffeine 2x220/65 mg vs Placebo; Test type: Other; p = 0.752, ANCOVA; geometric LS mean square = -0.07, 95% CI 2-sided [-0.49 to 0.35]
Statistical Analysis 10: Comparison: Naproxen Sodium/ Caffeine 220/65 mg vs Placebo; Test type: Other; p = 0.321, ANCOVA; geometric LS mean square = -0.21, 95% CI 2-sided [-0.63 to 0.21]

12. Secondary Outcome: Number of Participants With Certain Peak Pain Relief Score
Description: Number of participants with pain relief score 4, 3, 2, 1. The Peak Pain Relief Score refers to the highest level of pain relief a participant reported at any time point during the study period. It provides an overview of the maximum effectiveness of the treatment at any given point during the observation period using the Categorical Pain Relief Scale which measure the degree of pain relief using a scale from 0 to 4, in which 0 is no relief, 1 a little relief, 2 some relief, 3 a lot of relief and 4 complete relief. A high socre closer indicates significant pain relief and reflects the effectiveness of the analgesic treatment. A score closer to 0 indicates little to no pain relief and suggests limited treatment efficacy.
Time Frame: Up to 24 hours post-dose
Measure: Count of Participants; unit: Participants
Arm/Group | Naproxen Sodium/ Caffeine 220/65 mg | Naproxen Sodium/Caffeine 2x220/65 mg | Naproxen Sodium 220 mg | Caffeine 100 mg | Placebo
Number analyzed (Participants) | 147 | 148 | 147 | 50 | 49
Participants
  Pain relief score 4 | 31 | 47 | 36 | 15 | 15
  Pain relief score 3 | 101 | 85 | 102 | 31 | 29
  Pain relief score 2 | 14 | 15 | 9 | 4 | 5
  Pain relief score 1 | 1 | 1 | 0 | 0 | 0

13. Secondary Outcome: Cumulative Percent of Participants With 'at Least a 2-point PID' Over Time
Time Frame: Up to 24 hours post-dose
Measure: Number; unit: percentage
Arm/Group | Naproxen Sodium/ Caffeine 220/65 mg | Naproxen Sodium/Caffeine 2x220/65 mg | Naproxen Sodium 220 mg | Caffeine 100 mg | Placebo
Number analyzed (Participants) | 147 | 148 | 147 | 50 | 49
percentage
  0.5 hour post-dose | 50.3 | 62.8 | 60.5 | 32.0 | 18.4
  less or equal 1 hour | 78.2 | 86.5 | 86.4 | 40.0 | 26.5
  less or equal 1.5 hour | 87.1 | 94.6 | 92.5 | 46.0 | 40.8
  less or equal 2 hours | 92.5 | 98.0 | 94.6 | 64.0 | 71.4
  less or equal 3 hours | 98.0 | 99.3 | 98.0 | 86.0 | 87.8
  less or equal 4 hours | 98.6 | 99.3 | 99.3 | 94.0 | 95.9
  less or equal 5 hours | 98.6 | 99.3 | 99.3 | 98.0 | 98.0
  less or equal 6 hours | 99.3 | 99.3 | 99.3 | 100 | 98.0
  less or equal 7 hours | 99.3 | 99.3 | 99.3 | 100 | 98.0
  less or equal 8 hours | 99.3 | 99.3 | 100 | 100 | 98.0
  less or equal 9 hours | 99.3 | 99.3 | 100 | 100 | 98.0
  less or equal 10 hours | 99.3 | 99.3 | 100 | 100 | 98.0
  less or equal 11 hours | 99.3 | 99.3 | 100 | 100 | 98.0
  less or equal 12 hours | 100 | 99.3 | 100 | 100 | 98.0
  less or equal 14 hours | 100 | 99.3 | 100 | 100 | 98.0
  less or equal 16 hours | 100 | 99.3 | 100 | 100 | 98.0
  less or equal 18 hours | 100 | 99.3 | 100 | 100 | 98.0
  less or equal 20 hours | 100 | 99.3 | 100 | 100 | 98.0
  less or equal 22 hours | 100 | 99.3 | 100 | 100 | 98.0
  less or equal 24 hours | 100 | 99.3 | 100 | 100 | 98.0

14. Secondary Outcome: Global Assessment of Pain Relief of the Investigational Product
Description: Number of participants with overall rating poor, fair, good, very good, excellent 24 hour post-dose
Time Frame: 24 hours post-dose
Measure: Count of Participants; unit: Participants
Arm/Group | Naproxen Sodium/ Caffeine 220/65 mg | Naproxen Sodium/Caffeine 2x220/65 mg | Naproxen Sodium 220 mg | Caffeine 100 mg | Placebo
Number analyzed (Participants) | 147 | 146 | 147 | 50 | 47
Participants
  poor | 16 | 5 | 11 | 26 | 27
  fair | 10 | 12 | 12 | 10 | 5
  good | 35 | 23 | 38 | 8 | 3
  very good | 56 | 69 | 58 | 5 | 9
  excellent | 30 | 37 | 28 | 1 | 3

15. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of participants with at least one treatment emergent adverse event
Time Frame: Up to 5 days post-dose
Measure: Count of Participants; unit: Participants
Arm/Group | Naproxen Sodium/ Caffeine 220/65 mg | Naproxen Sodium/Caffeine 2x220/65 mg | Naproxen Sodium 220 mg | Caffeine 100 mg | Placebo
Number analyzed (Participants) | 147 | 148 | 147 | 50 | 49
Participants | 19 | 11 | 23 | 3 | 4

16. Secondary Outcome: Number of Participants With Significant Changes in Vital Signs Since Baseline
Time Frame: Up to 5 days post-dose
Measure: Number; unit: Participants
Arm/Group | Naproxen Sodium/ Caffeine 220/65 mg | Naproxen Sodium/Caffeine 2x220/65 mg | Naproxen Sodium 220 mg | Caffeine 100 mg | Placebo
Number analyzed (Participants) | 147 | 148 | 147 | 50 | 49
Participants
  Bradycardia | 1 | 1 | 0 | 0 | 0
  Tachycardia | 1 | 0 | 3 | 0 | 0
  Hypertension | 2 | 0 | 0 | 0 | 0
  Hypotension | 1 | 3 | 4 | 0 | 0

ADVERSE EVENTS:
Time Frame: All AEs and SAEs were collected from the signing of the ICF until last contact (follow-up visit at 2-5 days after discharge), an average of 5 days.
Arm/Group | Naproxen Sodium/ Caffeine 220/65 mg | Naproxen Sodium/Caffeine 2x220/65 mg | Placebo | Caffeine 100 mg | Naproxen Sodium 220 mg
All-Cause Mortality (participants affected / at risk) | 0/147 | 0/148 | 0/49 | 0/50 | 0/147
Serious Adverse Events (participants affected / at risk) | 0/147 | 0/148 | 0/49 | 0/50 | 0/147
Other Adverse Events (participants affected / at risk) | 19/147 | 11/148 | 4/49 | 3/50 | 23/147
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naproxen Sodium/ Caffeine 220/65 mg (N=147) | Naproxen Sodium/Caffeine 2x220/65 mg (N=148) | Placebo (N=49) | Caffeine 100 mg (N=50) | Naproxen Sodium 220 mg (N=147)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alveolar osteitis (Infections and infestations) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (4) | 2 (2) | 1 (1) | 0 (0) | 7 (7)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 0 (0) | 3 (3) | 1 (2) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 6 (7) | 0 (0) | 0 (0) | 5 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 9 (12)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2023-03-13): https://cdn.clinicaltrials.gov/large-docs/05/NCT05485805/Prot_006.pdf
  • Statistical Analysis Plan (2024-03-11): https://cdn.clinicaltrials.gov/large-docs/05/NCT05485805/SAP_007.pdf